CLINICAL TRIAL: NCT07027150
Title: Pulse Oximeter Validation Study for the Perin Health Patch
Status: Completed | Type: Observational
Sponsor: Perin Health Devices (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: PHD-25-002
Record Dates: First submitted 2025-05-23; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Hypoxia
Keywords: Hypoxia; Desaturation; Pulse Oximetry
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Healthy Volunteer: This cohort includes healthy adult volunteers aged 18-50 who undergo controlled hypoxemia testing to evaluate the performance of the Perin Health Patch, a chest-worn pulse oximeter. Each participant will be fitted with the Perin Health Patch and one or more FDA-cleared reference pulse oximeters. Under the supervision of trained clinicians, inspired oxygen concentrations will be adjusted to achieve stable oxygen saturation plateaus between 70% and 100%. Arterial blood samples will be collected and analyzed via co-oximetry to determine true functional SaO₂ values. Device performance will be assessed by comparing the SpO₂ readings from the Perin Health Patch with these reference values in accordance with ISO 80601-2-61.
  Interventions: Device: Chest Worn Pulse Oximeter

INTERVENTIONS:
Device: Chest Worn Pulse Oximeter — The Perin Health Patch is a non-invasive, chest-worn wearable device designed to continuously monitor physiological signals, including photoplethysmography (PPG), oxygen saturation (SpO₂), electrocardiography (ECG), and other health metrics. In this study, the device will be evaluated for its ability to accurately measure SpO₂ during controlled hypoxemia in healthy adult volunteers. The SpO₂ values recorded by the Perin Health Patch will be compared against arterial oxygen saturation values (SaO₂) obtained via co-oximetry, following the UCSF Hypoxia Lab protocol aligned with ISO 80601-2-61 standards.
  This device integrates PPG and ECG sensors into a single chest-applied unit, distinguishing it from conventional finger or earlobe pulse oximeters. The intervention in this study is limited to the application and use of the device for data collection under clinically controlled oxygen saturation conditions.

SUMMARY:
The goal of this clinical trial is to evaluate the accuracy of the Perin Health Patch, a chest-worn pulse oximeter, in healthy adult volunteers by comparing its measurements to arterial blood gas analysis during controlled hypoxemia. This study will help determine whether the device meets the performance requirements of ISO 80601-2-61 and FDA 510(k) for SpO₂ measurement accuracy.

The main questions it aims to answer is whether the Perin Health Patch meet the required accuracy performance (Arms ≤ 3.5%) across the full range of 70-100% SaO₂ as defined by ISO 80601-2-61.

Participants will be healthy adults aged 18 to 50 years old, representing a diverse range of skin tones (including ≥15% with Fitzpatrick V or VI). Inclusion criteria require general good health and no chronic medical conditions. Exclusion criteria include obesity, cardiopulmonary conditions, hemoglobinopathies, pregnancy, and other safety considerations.

Participants will:

* Undergo screening and informed consent, including skin tone assessment using colorimetry and spectrophotometry.
* Be instrumented with the Perin Health Patch and reference pulse oximeters on randomized fingers.
* Undergo placement of an arterial catheter by a trained physician.
* Be asked to breathe through a mouthpiece while inspired oxygen concentration is gradually reduced under physician control to generate multiple plateaus of hypoxemia (70-100% SaO₂).
* Provide up to 30 arterial blood samples at steady-state hypoxemia levels to determine functional SaO₂ via co-oximetry.
* Be continuously monitored for SpO₂, heart rate, ECG, respiratory rate, and blood pressure during the study.
* Return to normoxia, and have the arterial line removed with hemostasis confirmed before discharge.

This protocol, based on UCSF's standard hypoxia lab procedures, has been used in over 3000 subjects and is designed to meet or exceed requirements of ISO 80601-2-61, ISO 14155, and FDA 510(k) standards.

DETAILED DESCRIPTION:
This study is designed to evaluate the oxygen saturation measurement performance of the Perin Health Patch, a chest-worn pulse oximeter, during controlled hypoxemia in healthy adult volunteers. The study is conducted using UCSF's standard protocol for pulse oximeter performance evaluation, which has historically informed FDA and ISO standards (including ISO 80601-2-61). The Perin Health Patch integrates photoplethysmography (PPG) and other sensing modalities into a wearable form factor intended for clinical and non-clinical monitoring settings.

Participants will be enrolled to ensure demographic diversity, including representation across a wide spectrum of skin pigmentation, with a minimum of 15% of subjects having Fitzpatrick skin type V or VI. The study will control inspired gas concentrations to induce stable arterial oxygen saturation plateaus between 70% and 100%. These plateaus enable comparison of the device's displayed SpO₂ values to gold-standard SaO₂ values determined from arterial blood samples using co-oximetry.

SpO₂ readings from the Perin Health Patch will be collected concurrently with FDA-cleared reference pulse oximeters placed on contralateral or adjacent fingers. Readings at each plateau will be compared to SaO₂ to assess device accuracy and bias across the range of hypoxemia. The study will follow ISO 80601-2-61 methodology, including at least 200 paired data points from a minimum of 10 subjects. Averaging times and perfusion indices will be documented for all devices.

Data will be analyzed to determine root mean square error (Arms), bias, and standard deviation between device SpO₂ and co-oximeter SaO₂ readings. The results will be used to assess whether the Perin Health Patch meets regulatory performance requirements for oxygen saturation monitoring and to support future regulatory submissions.

This study does not involve randomization to different treatments or control arms. All participants undergo the same measurement protocol. No investigational treatments are administered. Safety protocols, including continuous vital sign monitoring and immediate availability of emergency medical care, are employed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* The subject is aged ≥18 and <50.
* The subject is in good general health with no evidence of any medical problems.
* The subject is fluent in both written and spoken English (we are actively working to expand access to this study to subjects who prefer other languages)
* The subject has provided informed consent and is willing to comply with the study procedures

Exclusion Criteria:

* The subject is obese (BMI>30).
* The subject has a known history of heart disease, lung disease, kidney or liver disease.
* Diagnosis of asthma, sleep apnea, or use of CPAP.
* Subject has diabetes.
* Subject has a clotting disorder.
* The subject a hemoglobinopathy or history of anemia, per subject report or the first blood sample, that in the opinion of the investigator, would make them unsuitable for study participation.
* The subject has any other serious systemic illness.
* The subject is a current smoker.
* Any injury, deformity, or abnormality at the sensor sites that in the opinion of the investigators' would interfere with the sensors working correctly.
* The subject has a history of fainting or vasovagal response.
* The subject has a history of sensitivity to local anesthesia.
* The subject has a diagnosis of Raynaud's disease.
* The subject has unacceptable collateral circulation based on an exam by the investigator (Allen's test).
* The subject is pregnant, lactating or trying to get pregnant.
* The subject is unable or unwilling to provide informed consent, or is unable or unwilling to comply with study procedures.
* The subject has any other condition, which in the opinion of the investigators' would make them unsuitable for the study.
* Subjects are screened for COVID 19 before coming in for testing. Fully vaccinated subjects are recruited for this study. Subjects will be asked if they have any symptoms related to COVID -19 and if they have any symptoms or are sick they cannot participate and a temperature will be taken before the study.
* The subject has recently been injected with methylene blue.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of healthy adult volunteers between the ages of 18 and 50 years, recruited to ensure adequate demographic and skin tone diversity. At least 15% of participants will have Fitzpatrick skin types V or VI. All participants must be in good general health, with no history of chronic cardiovascular, pulmonary, hematologic, renal, or hepatic conditions. Volunteers are excluded if they have a body mass index (BMI) greater than 30, are current smokers, or have any contraindications to arterial line placement or hypoxia exposure. Pregnant or lactating individuals are also excluded. All participants must provide informed consent and be fully vaccinated against COVID-19. The population is limited to English-speaking individuals due to current protocol constraints.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2025-05-27 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Accuracy of Perin Health Patch SpO₂ Measurements Compared to Arterial Blood Gas SaO₂ | During a single in-lab hypoxemia session lasting approximately 1 hour per participant
  The primary outcome is the accuracy of the oxygen saturation (SpO₂) values reported by the Perin Health Patch compared to functional arterial oxygen saturation (SaO₂) measured by co-oximetry from arterial blood samples. Accuracy will be assessed according to ISO 80601-2-61 standards using root-mean-square error (Arms), bias (mean difference), and standard deviation. Measurements will be collected at multiple stable plateaus of oxygen saturation induced by adjusting inspired gas concentrations in a controlled laboratory setting. Each comparison will be made at steady-state conditions, verified by reference pulse oximeters and end-tidal gas analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Hypoxia Lab, San Francisco, California, United States

DOCUMENTS (1):
  • Study Protocol (2024-10-24): https://cdn.clinicaltrials.gov/large-docs/50/NCT07027150/Prot_000.pdf